CLINICAL TRIAL: NCT03430271
Title: ENhancing Independence Using Group-based Community Interventions for Healthy AGing in Elders: The ENGAGE Pilot Study
Acronym: ENGAGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Collaborators: Somerville Council on Aging (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 11624
Record Dates: First submitted 2017-10-26; First posted 2018-02-12 (Actual); Last update posted 2018-02-14 (Actual); Status verified 2018-02

CONDITIONS: Mobility Limitation
MeSH Terms: conditions — Mobility Limitation

STUDY DESIGN:
Intervention Model Description: The ENGAGE Somerville Study is designed as a single blind, randomized-controlled, parallel-group pilot study. This study plans to enroll up to 50 participants to be randomized into the PA or health aging intervention.
Who Masked: Outcomes Assessor
Masking Description: The study assessor will be blinded to the treatment assignment. The study investigators and interventionists will not be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical Activity (PA) Intervention (Active Comparator)
  Interventions: Other: Physical Activity Intervention
- Health Education (HE) Intervention (Placebo Comparator)
  Interventions: Other: Healthy Aging Intervention

INTERVENTIONS:
Other: Physical Activity Intervention — Participants in this arm will complete exercise sessions 1 time per week for 24 weeks. An optional, second PA session will also be offered to PA participants. The exercise sessions will be multimodal and involve walking, lower extremity strengthening exercises, flexibility and balance training.
  Arms: Physical Activity (PA) Intervention
Other: Healthy Aging Intervention — Participants will attend health education workshops on topics of relevance to older adults. Workshops will be offered weekly in a group setting, and participants will be required to attend biweekly.
  Arms: Health Education (HE) Intervention

SUMMARY:
This study will be conducted to determine the safety and feasibility of translating a physical activity intervention (LIFE Study) into a community setting. Study outcomes include physical performance, safety, and feasibility of conducting the LIFE PA intervention in a community setting.

DETAILED DESCRIPTION:
Older adults who lose their mobility experience a poorer quality of life, are less likely to remain independent in the community and have higher rates of chronic disease, falls and mortality. Recent results from the Lifestyle Interventions and Independence for Elders (LIFE) study demonstrated that a structured program of physical activity (PA) reduced the onset of major mobility disability in at-risk older adults by up to 28% over a 2.6 year period. Despite the public health significance of this study, to-date no study has attempted to translate LIFE PA to broader populations of at-risk older adults in community-based settings. To address this knowledge gap, and to aid the design of a larger pragmatic trial of LIFE PA in community-based settings, the investigators conducted the ENhancing independence using Group-based community interventions for healthy AGing in Elders (ENGAGE) pilot study. The investigators examined the safety and feasibility of translating LIFE PA into the existing infrastructure of a community-based senior center. The investigators also explored the preliminary real-world effectiveness of PA on physical performance and several other important health related outcomes for older persons, including cognitive function, quality of life, depressive symptoms and frequency of falling.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females age ≥ 65 and ≤89 years
* Community dwelling
* Short Physical Performance Battery ≤ 9
* No participation in a structured physical activity program within the previous 3 months
* Willingness to be randomized and participate for 24 weeks
* Written permission from primary care physician
* Having obtained his/her informed consent

Exclusion Criteria:

* Acute or terminal illness
* Modified Mini-Mental State Examination Score <80(<76 if African American)*
* Myocardial Infarction in the previous 6 months
* Symptomatic coronary artery disease
* Upper or lower extremity fracture in the previous 6 months
* Resting blood pressure >180/100 mmHg
* Unable to communicate due to severe hearing loss or speech disorder
* Severe visual impairment that may preclude participation in the study assessments or interventions
* Non-English speaking

Ages: 65 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 59 (Actual)
Dates: Start 2015-05-12 (Actual); Primary Completion 2016-06-30 (Actual); Study Completion 2016-06-30 (Actual)

PRIMARY OUTCOMES:
This study will assess the safety of translating LIFE PA to a real-world community based setting by monitoring the occurrence of adverse events and serious adverse events. | 6 months
  Safety will be measured by the number of adverse events and serious adverse events. The investigators will compare the rates of adverse events and serious adverse events between the physical activity and healthy aging education intervention randomized arms.
This study will assess the feasibility of translating LIFE PA to a real-world community based setting with adequate PA adherence in the community by measuring intervention adherence and retention. | 6 months
  Intervention adherence is measured by percent attendance (number of visits attended/total number of scheduled visits). Successful adherence will be defined by an attendance rate of >60%. This will be used as an index of feasibility.

SECONDARY OUTCOMES:
Accelerometry | 6 months
  Accelerometry will objectively measure levels of physical activity intensity (light/moderate) and sedentary time. Accelerometry will be measured by GT3X+, Actigraph, Pensacola, FL. The actigraph will be worn for a 7-day period during waking hours during baseline and follow-up. This outcome measure will be assessed by the change in measurements between baseline and 24 weeks
Short physical performance battery (SPPB) test (an additional interim SPPB assessment will be conducted at week 12) | 6 months
  The SPPB test will be evaluated using a 4m gait speed test, chair stand test (consisting of five consecutive chair stands), and a balance test (measured by a side-by-side, semi-tandem, and full tandem stand). This test will assess the time to complete a 4m walk and a chair stand test, as well as the time each participant can hold the balance positions (up to 10 seconds). Time will be measured in minutes and seconds. This outcome measure will be assessed by the change in measurements between baseline and 24 weeks.
400 meter walk | 6 months
  The 400 meter walk will be a timed measurement of 10 laps around a 20 meter course or until the participant is unable to continue. Time will be measured in minutes and seconds. This outcome measure will be assessed by the change in measurements between baseline and 24 weeks.
Quality of Well-Being | 6 months
  This assessment will be measured using the Quality of Well-Being (QWB) Scale questionnaire. This scale provides a comprehensive measure of health-related quality of life that assesses health symptoms and functioning. The questionnaire is scored using a 0 to 1.0 scale (0 representing death, 1.0 representing asymptomatic full function). This outcome measure will be assessed by the change in measurements between baseline and 24 weeks.
Depressive symptoms | 6 months
  Depressive symptoms will be assessed using the Center for Epidemiologic Studies Depression Scale (CES-D), which is designed to measure depressive symptomology in the general population. The Scale consists of 20 questions, which are assigned a response score of 0, 1, 2 or 3 depending upon whether the item is worded positively or negatively. Possible range of total scores is 0 to 60, with the higher scores indicating the presence of more symptomatology. A cutoff score of 16 or greater reflects individuals at risk for clinical depression. This outcome measure will be assessed by the change in measurements between baseline and 24 weeks.
Cognitive performance | 6 months
  Cognitive performance will be assessed using the Digit Symbol Substitution Test (DSST). The DSST is a measure of attention and perceptual speed in which subjects are given a series of numbered symbols and then asked to draw the appropriate symbols below a list of random numbers. The score is the number of correctly made matches in 2 minutes. This outcome measure will be assessed by the change in measurements between baseline and 24 weeks.
Hand-Grip Strength | 6 months
  Grip strength will be measured in the dominant hand with a Jamar Handheld Dynamometer. Participants will be asked to perform a maximal isometric contraction. Strength will be measured in kilograms. This outcome measure will be assessed by the change in measurements between baseline and 24 weeks.
Nutrition Status | 6 months
  Nutrition Status will be assessed using the Mini Nutrition Assessment, Short Form (MNA-SF). The MNA-SF is a validated nutrition screening assessment tool that can identify geriatric patients age 65 and above who are malnourished or at risk of malnutrition. This outcome measure will be assessed by the change in measurements between baseline and 24 weeks.
Falls history | 6 months
  Participants will be asked about any recent falls they have experienced at each assessment visit and will be asked to record any falls that they experience throughout the trial on a calendar provided by the study interventionist. Falls history will be reported from baseline to 24 weeks.
Isometric Leg strength | 6 months
  Maximal isometric leg strength will be assessed using a portable electronic weight scale. Participants will be instructed to kick their leg as hard as possible three times on each leg. This outcome measure will be assessed by the change in measurements between baseline and 24 weeks.
Complex Walking Tasks (CWT's) | 6 months
  Subjects will be asked to walk on an even surface for 7 meters as fast as possible while remaining safe. They will then be asked to repeat the walk at their usual pace while simultaneously subtracting 3 from 50 and keep subtracting until the 7 meter walk is completed. The walk will be timed (measured in minutes with a stop watch and each subtraction will be recorded. This outcome measure will be assessed by the change in measurements between baseline and 24 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Kieran Reid, PhD, Principal Investigator — Tufts University
Locations (2):
- United States (2):
  - Jean Mayer Human Nutrition Research Center on Aging at Tufts University, Boston, Massachusetts
  - Somerville Council on Aging Holland Street Senior Center, Somerville, Massachusetts

REFERENCES:
- [Background] Gardener EA, Huppert FA, Guralnik JM, Melzer D. Middle-aged and mobility-limited: prevalence of disability and symptom attributions in a national survey. J Gen Intern Med. 2006 Oct;21(10):1091-6. doi: 10.1111/j.1525-1497.2006.00564.x. PMID 16970558
- [Background] Leveille SG, Guralnik JM, Ferrucci L, Langlois JA. Aging successfully until death in old age: opportunities for increasing active life expectancy. Am J Epidemiol. 1999 Apr 1;149(7):654-64. doi: 10.1093/oxfordjournals.aje.a009866. PMID 10192313
- [Background] Guralnik JM, Ferrucci L, Pieper CF, Leveille SG, Markides KS, Ostir GV, Studenski S, Berkman LF, Wallace RB. Lower extremity function and subsequent disability: consistency across studies, predictive models, and value of gait speed alone compared with the short physical performance battery. J Gerontol A Biol Sci Med Sci. 2000 Apr;55(4):M221-31. doi: 10.1093/gerona/55.4.m221. PMID 10811152
- [Background] Guralnik JM, Simonsick EM, Ferrucci L, Glynn RJ, Berkman LF, Blazer DG, Scherr PA, Wallace RB. A short physical performance battery assessing lower extremity function: association with self-reported disability and prediction of mortality and nursing home admission. J Gerontol. 1994 Mar;49(2):M85-94. doi: 10.1093/geronj/49.2.m85. PMID 8126356
- [Background] Hardy SE, Kang Y, Studenski SA, Degenholtz HB. Ability to walk 1/4 mile predicts subsequent disability, mortality, and health care costs. J Gen Intern Med. 2011 Feb;26(2):130-5. doi: 10.1007/s11606-010-1543-2. PMID 20972641
- [Background] Hubert HB, Bloch DA, Oehlert JW, Fries JF. Lifestyle habits and compression of morbidity. J Gerontol A Biol Sci Med Sci. 2002 Jun;57(6):M347-51. doi: 10.1093/gerona/57.6.m347. PMID 12023263
- [Background] LaCroix AZ, Guralnik JM, Berkman LF, Wallace RB, Satterfield S. Maintaining mobility in late life. II. Smoking, alcohol consumption, physical activity, and body mass index. Am J Epidemiol. 1993 Apr 15;137(8):858-69. doi: 10.1093/oxfordjournals.aje.a116747. PMID 8484377
- [Background] Stuck AE, Walthert JM, Nikolaus T, Bula CJ, Hohmann C, Beck JC. Risk factors for functional status decline in community-living elderly people: a systematic literature review. Soc Sci Med. 1999 Feb;48(4):445-69. doi: 10.1016/s0277-9536(98)00370-0. PMID 10075171
- [Background] Buchner DM, Beresford SA, Larson EB, LaCroix AZ, Wagner EH. Effects of physical activity on health status in older adults. II. Intervention studies. Annu Rev Public Health. 1992;13:469-88. doi: 10.1146/annurev.pu.13.050192.002345. PMID 1599599
- [Background] Dolansky MA, Moore SM. Effects of cardiac rehabilitation on the recovery outcomes of older adults after coronary artery bypass surgery. J Cardiopulm Rehabil. 2004 Jul-Aug;24(4):236-44. doi: 10.1097/00008483-200407000-00005. PMID 15286528
- [Background] Messier SP, Royer TD, Craven TE, O'Toole ML, Burns R, Ettinger WH Jr. Long-term exercise and its effect on balance in older, osteoarthritic adults: results from the Fitness, Arthritis, and Seniors Trial (FAST). J Am Geriatr Soc. 2000 Feb;48(2):131-8. doi: 10.1111/j.1532-5415.2000.tb03903.x. PMID 10682941
- [Background] Ades PA, Ballor DL, Ashikaga T, Utton JL, Nair KS. Weight training improves walking endurance in healthy elderly persons. Ann Intern Med. 1996 Mar 15;124(6):568-72. doi: 10.7326/0003-4819-124-6-199603150-00005. PMID 8597320
- [Background] Fielding RA, Rejeski WJ, Blair S, Church T, Espeland MA, Gill TM, Guralnik JM, Hsu FC, Katula J, King AC, Kritchevsky SB, McDermott MM, Miller ME, Nayfield S, Newman AB, Williamson JD, Bonds D, Romashkan S, Hadley E, Pahor M; LIFE Research Group. The Lifestyle Interventions and Independence for Elders Study: design and methods. J Gerontol A Biol Sci Med Sci. 2011 Nov;66(11):1226-37. doi: 10.1093/gerona/glr123. Epub 2011 Aug 8. PMID 21825283
- [Background] Pahor M, Guralnik JM, Ambrosius WT, Blair S, Bonds DE, Church TS, Espeland MA, Fielding RA, Gill TM, Groessl EJ, King AC, Kritchevsky SB, Manini TM, McDermott MM, Miller ME, Newman AB, Rejeski WJ, Sink KM, Williamson JD; LIFE study investigators. Effect of structured physical activity on prevention of major mobility disability in older adults: the LIFE study randomized clinical trial. JAMA. 2014 Jun 18;311(23):2387-96. doi: 10.1001/jama.2014.5616. PMID 24866862
- [Background] Teng EL, Chui HC. The Modified Mini-Mental State (3MS) examination. J Clin Psychiatry. 1987 Aug;48(8):314-8. PMID 3611032
- [Background] Choi L, Liu Z, Matthews CE, Buchowski MS. Validation of accelerometer wear and nonwear time classification algorithm. Med Sci Sports Exerc. 2011 Feb;43(2):357-64. doi: 10.1249/MSS.0b013e3181ed61a3. PMID 20581716
- [Background] Guralnik JM, Ferrucci L, Simonsick EM, Salive ME, Wallace RB. Lower-extremity function in persons over the age of 70 years as a predictor of subsequent disability. N Engl J Med. 1995 Mar 2;332(9):556-61. doi: 10.1056/NEJM199503023320902. PMID 7838189
- [Background] Newman AB, Simonsick EM, Naydeck BL, Boudreau RM, Kritchevsky SB, Nevitt MC, Pahor M, Satterfield S, Brach JS, Studenski SA, Harris TB. Association of long-distance corridor walk performance with mortality, cardiovascular disease, mobility limitation, and disability. JAMA. 2006 May 3;295(17):2018-26. doi: 10.1001/jama.295.17.2018. PMID 16670410
- [Background] Rantanen T, Guralnik JM, Foley D, Masaki K, Leveille S, Curb JD, White L. Midlife hand grip strength as a predictor of old age disability. JAMA. 1999 Feb 10;281(6):558-60. doi: 10.1001/jama.281.6.558. PMID 10022113
- [Background] Rantanen T, Harris T, Leveille SG, Visser M, Foley D, Masaki K, Guralnik JM. Muscle strength and body mass index as long-term predictors of mortality in initially healthy men. J Gerontol A Biol Sci Med Sci. 2000 Mar;55(3):M168-73. doi: 10.1093/gerona/55.3.m168. PMID 10795731
- [Background] Sherrington C, Lord SR. Reliability of simple portable tests of physical performance in older people after hip fracture. Clin Rehabil. 2005 Aug;19(5):496-504. doi: 10.1191/0269215505cr833oa. PMID 16119405
- [Background] Sink KM, Espeland MA, Rushing J, Castro CM, Church TS, Cohen R, Gill TM, Henkin L, Jennings JM, Kerwin DR, Manini TM, Myers V, Pahor M, Reid KF, Woolard N, Rapp SR, Williamson JD; LIFE Investigators. The LIFE Cognition Study: design and baseline characteristics. Clin Interv Aging. 2014 Aug 27;9:1425-36. doi: 10.2147/CIA.S65381. eCollection 2014. PMID 25210447
- [Background] Salthouse TA. The role of memory in the age decline in digit-symbol substitution performance. J Gerontol. 1978 Mar;33(2):232-8. doi: 10.1093/geronj/33.2.232. PMID 637915
- [Background] Kaplan RM, Ganiats TG, Sieber WJ, Anderson JP. The Quality of Well-Being Scale: critical similarities and differences with SF-36. Int J Qual Health Care. 1998 Dec;10(6):509-20. doi: 10.1093/intqhc/10.6.509. PMID 9928590
- [Background] Kaiser MJ, Bauer JM, Ramsch C, Uter W, Guigoz Y, Cederholm T, Thomas DR, Anthony P, Charlton KE, Maggio M, Tsai AC, Grathwohl D, Vellas B, Sieber CC; MNA-International Group. Validation of the Mini Nutritional Assessment short-form (MNA-SF): a practical tool for identification of nutritional status. J Nutr Health Aging. 2009 Nov;13(9):782-8. doi: 10.1007/s12603-009-0214-7. PMID 19812868
- [Background] Delbaere K, Close JC, Mikolaizak AS, Sachdev PS, Brodaty H, Lord SR. The Falls Efficacy Scale International (FES-I). A comprehensive longitudinal validation study. Age Ageing. 2010 Mar;39(2):210-6. doi: 10.1093/ageing/afp225. Epub 2010 Jan 8. PMID 20061508
- [Background] Yardley L, Beyer N, Hauer K, Kempen G, Piot-Ziegler C, Todd C. Development and initial validation of the Falls Efficacy Scale-International (FES-I). Age Ageing. 2005 Nov;34(6):614-9. doi: 10.1093/ageing/afi196. PMID 16267188